CLINICAL TRIAL: NCT04874766
Title: The Effects of Wearing a Face Mask on Exercise Tolerance in Children's Hockey During the COVID-19 Pandemic
Brief Title: The Effects of Wearing a Face Mask During Exercise in Youth Hockey Players During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2701
Record Dates: First submitted 2021-04-23; First posted 2021-05-06 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participant will be blinded by wearing a sham mask during the "no mask" condition (i.e. they will wear a surgical mask with the covering for the mouth and nose cut out). The individual who will statistically analyze the data will be blinded to conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical face mask (Experimental): Simulated hockey period with 2x20s Wingate tests; progressive-intensity on-ice sprint test while wearing a surgical mask
  Interventions: Other: Wingate exercise test and on-ice testing while wearing a face mask
- Sham face mask (Sham Comparator): Simulated hockey period with 2x20s Wingate tests; progressive-intensity on-ice sprint test while wearing a sham mask
  Interventions: Other: Wingate exercise test and on-ice testing while wearing a sham face mask

INTERVENTIONS:
Other: Wingate exercise test and on-ice testing while wearing a face mask — Power output during 2 x 20s Wingate cycle tests and total distance during an on-ice skating test while wearing a face mask
  Arms: Surgical face mask
Other: Wingate exercise test and on-ice testing while wearing a sham face mask — Power output during 2 x 20s Wingate cycle tests and total distance during an on-ice skating test while wearing a face mask
  Arms: Sham face mask

SUMMARY:
There is concern that wearing a face mask during COVID will affect oxygen uptake, especially during intense exercise. COVID transmission is especially prevalent in sports such as hockey, where there is close contact between players and arena ventilation is poor. This study will assess the effect of wearing a surgical face mask on simulated hockey performance and blood and muscle oxygenation during cycling exercise.

DETAILED DESCRIPTION:
The sport of ice hockey involves close contact between players in poorly ventilated arenas. This increases susceptibility for transmission of viruses, such as COVID-19. Face masks can reduce the risk of virus transmission; however, there is concern that wearing a face mask during exercise will reduce oxygen uptake or increase carbon dioxide re-breathing, which can result in low blood oxygen levels, reduced oxygen delivery to muscle and reduced exercise capacity. The purpose of the study is to determine the effect of wearing a surgical face mask during exercise that simulates ice hockey play on exercise performance and blood and muscle oxygenation in boys and girls. Twelve boys and twelve girls (age 9-14y) who are experienced playing hockey, will take part in this randomized cross-over study that will assess exercise performance, blood oxygenation (i.e. pulse oximetry) and muscle oxygenation (with near infrared spectroscopy) during an exercise test on a cycle ergometer with workloads and work to rest intervals that simulates hockey performance. Participants will also be tested for repeated-sprint performance on ice while wearing full hockey equipment. The conditions include no mask (a "sham" mask) and a surgical mask. Outcome variables include power output during the cycle ergometer testing, skating distance during the on-ice test, rating of perceived exertion, blood oxygen saturation levels, and oxygenated, deoxygenated, and total hemoglobin at the quadriceps muscle.

ELIGIBILITY:
Inclusion Criteria:

* Experience playing ice-hockey

Exclusion Criteria:

* Contra-indications to exercise as identified by a screening questionnaire (the "Get Active Questionnaire")

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in average power output | Up to 40 seconds
  Average power output in Watts during two 20 second Wingate tests

SECONDARY OUTCOMES:
Change from baseline in peak power output | Up to 40 seconds
  Peak power output in Watts during two 20 second Wingate tests
Change from baseline in on-ice sprint testing distance | Up to 12 minutes
  Distance in meters covered during a repeated 20-meter sprint test that progressively increases in speed
Change from baseline in blood oxygen saturation | Up to 40 minutes
  Blood oxygen saturation (%) determined by pulse oximetry
Change from baseline in quadriceps tissue oxygenation index | Up to 40 minutes
  Tissue oxygenation index (oxygenated hemoglobin/total hemoglobin) as measured by near infra-red spectroscopy
Change from baseline in rating of perceived exertion | Up to 40 minutes
  Rating of perceived exertion on a scale of 1-10 (Modified Borg Scale), a higher score indicates a greater perceived exertion
Change from baseline in heart rate | Up to 40 minutes
  Heart rate (beats per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, Ph.D., Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shaw KA, Butcher S, Ko JB, Absher A, Gordon J, Tkachuk C, Zello GA, Chilibeck PD. Wearing a Surgical Face Mask Has Minimal Effect on Performance and Physiological Measures during High-Intensity Exercise in Youth Ice-Hockey Players: A Randomized Cross-Over Trial. Int J Environ Res Public Health. 2021 Oct 14;18(20):10766. doi: 10.3390/ijerph182010766. PMID 34682512